CLINICAL TRIAL: NCT00155675
Title: Clinical Effect of Traditional Chinese Medicine - "Gusuibu"
Brief Title: Pseudodrynaria Coronana (Wall) Ching
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Sheng Chang Pharmaceutical (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 900505; CCMP90-RD-114
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

INTERVENTIONS:
Drug: GUSUIBU

SUMMARY:
The Study to evaluate the clinical effect of "Gusuibu" lasts for 3 years. It aims to evaluate its effect on bone density of postmenopausal osteoporosis. Besides, its effects on the liver, kidney and the hematological influence will be evaluated, too.

DETAILED DESCRIPTION:
Research of the this traditional chinese medicine clinucal, Gusuibu, curative effect is plan three years time. The entire studyaims to evaluated the effect of the traditional chinese medicine on postmenpausal osteoporosis as well as the possible side effects on the experimental animal and the human body. All subjects were postmenopausal woman with established osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal osteoporosis

Exclusion Criteria:

* Insulin dependent diabetes

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2000-01; Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
one year

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hwa-Chang, M.D, Study Chair — National Taiwan University Medical Center
Locations (1):
- National Taiwan University Medical Center, Taipei, 7, Chung-Shan S. Road, Taiwan